CLINICAL TRIAL: NCT06861413
Title: A Phase 1, Open-label, Randomized, Parallel Study to Evaluate the Relative Bioavailability of a Tablet Formulation of VX-828 in Healthy Adult Subjects
Brief Title: A Phase 1 Study to Evaluate the Relative Bioavailability of a VX-828 Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX25-828-002
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): Participants will be randomized to receive a single dose of VX-828 suspension.
  Interventions: Drug: VX-828
- Cohort 2 (Experimental): Participants will be randomized to receive a single dose of VX-828 tablets.
  Interventions: Drug: VX-828

INTERVENTIONS:
Drug: VX-828 — Tablets for Oral Administration.
  Arms: Cohort 2
Drug: VX-828 — Suspension for Oral Administration.
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of a VX-828 tablet formulation compared to a suspension and evaluate its safety and tolerability.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per square meter (kg/m^2)
* A total body weight of more than (>) 50 Kg
* Nonsmoker or ex-smoker for at least 3 months before screening
* Participants of non-childbearing potential

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve from the Time of dosing to the Last Measurable Concentration (AUC0-tlast) of VX-828 in Plasma | From Day 1 up to Day 24
Maximum Observed Concentration (Cmax) of VX-828 in Plasma | From Day 1 up to Day 24

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 36)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Tempe, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing